CLINICAL TRIAL: NCT02241122
Title: Improved Prostate Cancer Diagnosis - Combination of Magnetic Resonance Imaging Targeted Biopsies and Biomarkers (Multi-institutional Study)
Brief Title: MRI and Biomarkers in Prostate Cancer
Acronym: Multi-IMPROD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 72/1801/2014
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; PSA; MRI; biopsy; biomarker
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI guided prostate biopsy (Experimental): prostate biopsy after MR-imaging
  Interventions: Procedure: prostate biopsy

INTERVENTIONS:
Procedure: prostate biopsy

SUMMARY:
Prostate cancer has been the most common neoplastic disease in men in Finland over the last ten years. Prostate-specific antigen (PSA) plays an important role in screening of prostate cancer. However, PSA has a limited sensitivity and specificity for prostate cancer detection. Commonly, the diagnosis of prostate cancer is done by transrectal ultrasonography (TRUS) guided biopsy. Because of the low accuracy of TRUS a systematic biopsy is usually performed instead of targeted TRUS biopsy. As biopsy carries a significant risk of complications, there is an increasing interest in developing more accurate non-invasive imaging modalities.

This prospective multi-institutional study will enroll 400 men with clinical suspicion of prostate cancer due to higher serum level of PSA than 2.5 ng/ml and/or abnormal digital rectal examination. Anatomical magnetic resonance imaging (MRI) and diffusion weighted imaging (DWI) at 1.5/3 Tesla (T) magnetic field using surface coils will be used to non-invasively predict the presence or absence of prostate cancer. Targeted TRUS guided biopsy based on MRI findings will be performed in addition to routine twelve core TRUS biopsy. Moreover, selected serum and urine biomarkers as well as biomarkers extracted from fresh biopsy sample will be collected and correlated with the presence or absence of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 85 years
* Clinical suspicion of prostate cancer, based on: serum level of PSA from 2,5 ng/ml to 20 ng/ml in two following measurements and/or abnormal digital rectal examination
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient must sign the appropriate Ethics Committee (EC) approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* previous prostate biopsies within 6 months
* previous diagnosis of prostate carcinoma
* previous prostate surgeries, e.g. TURP (transurethral prostatic resection)
* symptomatic of acute prostatitis
* contraindications for MRI (cardiac pacemaker, intracranial clips etc)
* uncontrolled serious infection
* claustrophobia
* hip replacement surgery or other metal implants in the pelvic area

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-11 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of biparametric MRI (T2wi+DWI) in prostate cancer diagnosis | 18 months
  Biparametric MRI (T2wi+DWI) is performed in patients with a clinical suspicion of prostate cancer (elevated PSA and/or abnormal DRE). The accuracy will be determined using the results from transrectal ultrasound guided biopsies.

SECONDARY OUTCOMES:
Diagnostic accuracy of selected tissue, urine, and blood biomarkers for prostate cancer diagnosis | 18 months
  Accuracy of selected tissue, urine, and blood biomarkers for prostate cancer diagnosis will be evaluated.
  Gene expression profile of selected genes will be compared between cancer and non-cancer cases to investage optimal gene expression panels for prostate cancer risk prediction. Similarly serum and urine marker profiles are compared between cancer and non-cancer cases

OTHER OUTCOMES:
Evaluation of bacterial strains | 18 months
  The bacterial resistance towards antibiotics is evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Boström, MD, PhD, Principal Investigator — Department of Urology, University of Turku and Turku University Hospital
Locations (5):
- Finland (5):
  - Department of Urology, Helsinki University Hospital, Helsinki
  - Department of Urology, Kuopio University Hospital, Kuopio
  - Department of Urology, Pori Central Hospital, Pori
  - Department of Urology, Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

REFERENCES:
- [Background] Jambor I, Kahkonen E, Taimen P, Merisaari H, Saunavaara J, Alanen K, Obsitnik B, Minn H, Lehotska V, Aronen HJ. Prebiopsy multiparametric 3T prostate MRI in patients with elevated PSA, normal digital rectal examination, and no previous biopsy. J Magn Reson Imaging. 2015 May;41(5):1394-404. doi: 10.1002/jmri.24682. Epub 2014 Jun 23. PMID 24956412
- [Derived] Perez IM, Jambor I, Kauko T, Verho J, Ettala O, Falagario U, Merisaari H, Kiviniemi A, Taimen P, Syvanen KT, Knaapila J, Seppanen M, Rannikko A, Riikonen J, Kallajoki M, Mirtti T, Lamminen T, Saunavaara J, Pahikkala T, Bostrom PJ, Aronen HJ. Qualitative and Quantitative Reporting of a Unique Biparametric MRI: Towards Biparametric MRI-Based Nomograms for Prediction of Prostate Biopsy Outcome in Men With a Clinical Suspicion of Prostate Cancer (IMPROD and MULTI-IMPROD Trials). J Magn Reson Imaging. 2020 May;51(5):1556-1567. doi: 10.1002/jmri.26975. Epub 2019 Nov 21. PMID 31750988
- [Derived] Jambor I, Verho J, Ettala O, Knaapila J, Taimen P, Syvanen KT, Kiviniemi A, Kahkonen E, Perez IM, Seppanen M, Rannikko A, Oksanen O, Riikonen J, Vimpeli SM, Kauko T, Merisaari H, Kallajoki M, Mirtti T, Lamminen T, Saunavaara J, Aronen HJ, Bostrom PJ. Validation of IMPROD biparametric MRI in men with clinically suspected prostate cancer: A prospective multi-institutional trial. PLoS Med. 2019 Jun 3;16(6):e1002813. doi: 10.1371/journal.pmed.1002813. eCollection 2019 Jun. PMID 31158230
- [Derived] Knaapila J, Kallio H, Hakanen AJ, Syvanen K, Ettala O, Kahkonen E, Lamminen T, Seppanen M, Jambor I, Rannikko A, Riikonen J, Munukka E, Eerola E, Gunell M, Bostrom PJ. Antibiotic susceptibility of intestinal Escherichia coli in men undergoing transrectal prostate biopsies: a prospective, registered, multicentre study. BJU Int. 2018 Aug;122(2):203-210. doi: 10.1111/bju.14198. Epub 2018 Apr 6. PMID 29533507
- [Derived] Knaapila J, Gunell M, Syvanen K, Ettala O, Kahkonen E, Lamminen T, Seppanen M, Jambor I, Rannikko A, Riikonen J, Munukka E, Eerola E, Hakanen AJ, Bostrom PJ. Prevalence of Complications Leading to a Health Care Contact After Transrectal Prostate Biopsies: A Prospective, Controlled, Multicenter Study Based on a Selected Study Cohort. Eur Urol Focus. 2019 May;5(3):443-448. doi: 10.1016/j.euf.2017.12.001. Epub 2017 Dec 20. PMID 29275146